CLINICAL TRIAL: NCT00661466
Title: A Phase II, Randomized, Single-dose, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety and Pharmacokinetic Profile of the CollaRx Bupivacaine Implant in Patients After Gastrointestinal Surgery
Brief Title: Efficacy and Safety of A Collagen Bupivacaine Implant in Patients After Gastrointestinal Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INN-CB-004
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative
Keywords: Gastrointestinal surgery; Post operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Either three or four 5x5-cm bupivacaine sponges implanted at 2 sites within the surgical field (1) over the abdominal viscera and under the fascia prior to closing the fascia and (2) in the subcutaneous tissue just under the skin incision.
  Interventions: Drug: Bupivacaine Collagen Sponge
- 2 (Placebo Comparator): Either three or four 5x5-cm placebo sponges implanted at 2 sites within the surgical field (1) over the abdominal viscera and under the fascia prior to closing the fascia and (2) in the subcutaneous tissue just under the skin incision.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine Collagen Sponge
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the CollaRx Bupivacaine Implant (bupivacaine sponge) is safe and effective in reducing the amount of narcotic pain medication needed to control pain during the first 24 hours after gastrointestinal (GI) surgery.

DETAILED DESCRIPTION:
Gastrointestinal (GI) surgery encompasses a range of surgical procedures that involve abdominal incision. Gastrointestinal surgery may be performed to treat an abdominal aortic aneurysm, ulcerative colitis, Crohn's disease, gallbladder disease, bile duct disease and morbid obesity. Although less invasive laparoscopic procedures are performed when warranted, open abdominal surgery is required for certain indications and for more complicated or advanced cases.

Bupivacaine is a local anesthetic (pain medicine) that has an established safety profile. Collagen is a protein that is found in all mammals. The CollaRx Bupivacaine implant is a thin flat sponge made out of collagen that comes for cow tendons and contains bupivacaine. When inserted into a surgical site, the collagen breaks down and bupivacaine is released at the site but very little is absorbed into the blood stream. The high levels of bupivacaine at the surgical site may result in less pain for several days after surgery.

This study will compare the amount of narcotic pain medication required after surgery in patients who receive the CollaRx Bupivacaine implant or a plain collagen sponge.

ELIGIBILITY:
Inclusion Criteria:

* Must be a man or woman who is ≥ 18 and ≤ 75 years of age.
* Has a body mass index (BMI) > 19 and < 40 kg/m2.
* Has a planned elective surgery that requires a vertical or transverse abdominal incision (including but not limited to abdominal aortic aneurysm repair, cholecystectomy and simple bowel resection) to be performed according to standard surgical technique under general anesthesia.
* Has a risk classification of I, II or III according to the American Society of Anesthesiologists (ASA)
* If female, is nonpregnant (negative pregnancy test at Screening and Day 0 before surgery) and nonlactating.
* If female, is either not of childbearing potential or practicing a defined medically acceptable method of birth control and agrees to continue with the regimen throughout the study.
* Is free of other physical or mental conditions that, in the opinion of the Investigator, may confound quantification of postoperative pain resulting from the surgery.
* Has the ability and willingness to comply with the study procedures and the use of the pain scales; is deemed capable of operating a PCA device; and is able to communicate meaningfully with the study staff.
* Must voluntarily sign and date an informed consent form (ICF) that is approved by an IRB prior to the conduct of any study specific procedures.
* Must be able to fluently speak and understand English and be able to provide meaningful written informed consent for the study.

Exclusion Criteria:

* Has known hypersensitivity to amide local anesthetics, opioids or bovine products, or to inactive ingredients of the test article.
* Has 1 of the following surgical procedures planned: total abdominal hysterectomy, omentectomy or surgical procedure for staging cancer.
* Requires the use of Seprafilm® or other absorbable adhesion barriers for the GI surgery.

Requires any additional surgical procedures either related or unrelated to the GI surgery during the same hospitalization.

* Is required to receive neuraxial (spinal or epidural) opioid analgesics during the study.
* Has cardiac arrhythmia or atrioventricular (AV) conduction disorders.
* Concomitantly uses antiarrhythmics (eg, amiodarone), propranolol or strong/moderate cytochrome P450 (CYP) 3A4 inhibitors or inducers (eg, macrolide antibiotics and grapefruit juice).
* Has used long acting analgesics within 24 hours of surgery. Short acting analgesics such as acetaminophen may be used on the day of surgery but are subject to preoperative restrictions for oral intake.
* Has used aspirin or aspirin containing products within 7 days of surgery. Aspirin at a dose of ≤ 325 mg is allowed for cardiovascular prophylaxis if the patient has been on a stable dose regimen for ≥ 30 days prior to Screening.
* Has undergone another major surgery within 3 months of the GI surgery.
* Has known or suspected history of alcohol or drug abuse or misuse within 3 years of Screening or evidence of tolerance or physical dependency on opioid analgesics or sedative hypnotic medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-07-24; Primary Completion 2009-01-10 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Albany Medical Center Hospital, Albany, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated due to poor recruitment
Groups:
- 5x5-cm Bupivacaine Sponges: Either three or four 5x5-cm bupivacaine sponges implanted at 2 sites within the surgical field (1) over the abdominal viscera and under the fascia prior to closing the fascia and (2) in the subcutaneous tissue just under the skin incision.
  Bupivacaine Collagen Sponge
- 5x5-cm Placebo Sponges: Either three or four 5x5-cm placebo sponges implanted at 2 sites within the surgical field (1) over the abdominal viscera and under the fascia prior to closing the fascia and (2) in the subcutaneous tissue just under the skin incision.
  Placebo: placebo
Period: Overall Study
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Started | 4 (Participants) | 3 (Participants)
Completed | 4 (Participants) | 3 (Participants)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Total Amount of Opioid Rescue Analgesia Used
Description: Study Terminated early due to very poor study enrollment. Target recruitment not met. Primary outcome not measured - planned statistical analyses was not performed.
Time Frame: 0 to 24 hours postoperatively
Population: Study Terminated early due to very poor study enrollment. Target recruitment not met. Primary outcome not measured - planned statistical analyses was not performed.
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Total Amount of Opioid Rescue Analgesia Used
Description: Study Terminated Early - Secondary end point not measured - not done - Study Terminated early due to very poor study enrollment. Target recruitment not met. Primary outcome not measured - planned statistical analyses was not performed.
Time Frame: 0 to 48 hours postoperatively
Population: Study Terminated Early - Secondary end point not measured - not done
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Total Amount of Opioid Rescue Analgesia Used
Description: as for outcome 2
Time Frame: 0 to 72 hours postoperatively
Population: Study Terminated Early - Secondary end point not measured - not done - Study Terminated early due to very poor study enrollment. Target recruitment not met. Primary outcome not measured - planned statistical analyses was not performed.
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain Intensity Rating on the Visual Analogue Scale (VAS)
Description: as for outcome 2
Time Frame: 1, 1.5, 2, 3, 4, 5, 6, 24, 48 and 72 hours after Time 0
Population: as for outcome 3
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain Intensity Rating on a 4-point Scale
Description: Study Terminated Early - Secondary end point not measured - not done
Time Frame: At 1, 1.5, 2, 3, 6, 9, 12, 18, 24, 36, 48 and 72 hours postoperatively
Population: Study Terminated Early - Secondary end point not measured - not done
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pain Relief Rating on a 5-point Scale
Description: as for outcome 2
Time Frame: At 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 24, 48 and 72 hours after Time 0
Population: as for outcome 3
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Patient Global Evaluation of Study Treatment on a 5-point Scale
Description: Study Terminated Early - Secondary end point not measured - not done
Time Frame: At 72 hours after time 0
Population: Study Terminated Early - Secondary end point not measured - not done
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to First Use of Opioid Rescue Analgesia
Description: as for outcome 2
Time Frame: actual time from time 0
Population: as for outcome 3
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pharmacokinetic Parameters
Description: as for outcome 2
Time Frame: 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours postoperatively
Population: as for outcome 3
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: The Incidence of Treatment-emergent Adverse Events
Description: as for outcome 2
Time Frame: Through 30 days after surgery
Population: as for outcome 3
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Changes in Vital Sign Measurements
Description: as for outcome 2
Time Frame: Through 72 hours post insertion
Population: as for outcome 3
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Information regarding AEs was collected from the time of hospital admission through Day 30. Normal postoperative sequelae were not considered to be AEs unless they occurred in a more severe form, as judged by the investigator. Information on AEs was also collected during the Day 8 and Day 30 follow-up calls.
Arm/Group | 5x5-cm Bupivacaine Sponges | 5x5-cm Placebo Sponges
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5x5-cm Bupivacaine Sponges (N=4) | 5x5-cm Placebo Sponges (N=3)
hypotension (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5x5-cm Bupivacaine Sponges (N=4) | 5x5-cm Placebo Sponges (N=3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Arm Pain -IV Site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Polyuria (Gastrointestinal disorders) | 0 (0) | 1 (1)
Marcaine Sensitivity (Product Issues) | 1 (1) | 0 (0)
Prolonged QT interval (Cardiac disorders) | 1 (1) | 0 (0)
shivering (General disorders) | 0 (0) | 1 (1)
elevated temperature (General disorders) | 1 (1) | 0 (0)
surgical wound seroma (Surgical and medical procedures) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No